CLINICAL TRIAL: NCT07368621
Title: Effectiveness of Connective Tissue Graft With and Without Leukocyte Platelet Rich Fibrin on Peri-implant Soft Tissue Thickness Around Delayed Implants in Patients With Thin Gingival Phenotype: A Randomized Controlled Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: British University In Egypt (Other)
Responsible Party: Principal Investigator, Rania hesham, Demonstrator, British University In Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23-051
Record Dates: First submitted 2026-01-20; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Soft Tissue Thickness Around Delayed Implants in Patients With Thin Gingival Phenotype
Keywords: CTG; L-Prf; Soft tissue thickness

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Biostatican
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): Connective tissue graft (CTG)
  Interventions: Procedure: Connective tissue graft(CTG)
- Test group (Active Comparator): Connective tissue graft (CTG) + leukocyte platelet-rich fibrin (L-PRF)
  Interventions: Procedure: Connective tissue graft (CTG) + leukocyte platelet-rich fibrin (L-PRF)

INTERVENTIONS:
Procedure: Connective tissue graft(CTG) — A harvested connective tissue graft will be placed in the prepared muco-periosteal flap around the implant. The graft will be adapted and secured in place using horizontal matrices.
  Arms: Control group
Procedure: Connective tissue graft (CTG) + leukocyte platelet-rich fibrin (L-PRF) — To prepare the L-PRF, a 10 ml of blood will be drawn from the antecubital vein of the patient's right or left arm and will be transferred to the free anticoagulant test-tube. The blood sample will be immediately centrifuged at 2700 rpm for 12 minutes33. L-PRF will be applied over the connective tissue graft in the prepared mucoperiosteal flap around the implant34. Then the graft will be secured with horizontal mattresses with an absorbable vicryl 6-0. A non-absorbable prolene suture will be used to approximate the flap.
  Arms: Test group

SUMMARY:
A stable soft and hard tissues around Osseo-integrated implants are very crucial. Soft tissue thickness around implants is crucial as it prevents peri-implant bone loss and enhance the esthetic outcomes. The treatment of thin tissue phenotype should be improved as the thin tissue phenotype will lead to plaque accumulation. There are some techniques that can increase the thickness of the peri-implant mucosa including connective tissue graft, platelet- rich fibrin and xenogeneic collagen matrix .Leukocyte and Platelet rich fibrin is a second generation platelet concentrate that was introduced by choukroun et al in 2001 after platelet rich plasma. PRF is the first source of autogenous blood derived growth factors harvested without the use of anticoagulants5. It contains various growth factors that are believed to contribute to periodontal regeneration. It promotes neovascularization and accelerated wound closing

DETAILED DESCRIPTION:
Soft tissue thickness around implants is crucial as it prevents peri-implant bone loss and enhance the esthetic outcomes. The critical amount of soft tissue thickness on the buccal aspect of implants has been determined to be 2mm. Thick mucosal tissue often has better esthetic outcomes as it creates better tissue contour, mask the metal abutment and creating papilla after prosthesis fabrication. The difference in the amount of bone remodeling is related to the difference in mucosal tissue thickness, which is believed to be the result of supracrestal tissue height establishment. Presence of thin gingival phenotype around dental implant increases the prevalence of peri-implantitis and peri-implant mucositis. Thin gingival phenotype and inadequate keratinized mucosa width lead to greater food impaction compared with thick gingival phenotype and adequate keratinized mucosa. Patients with thin gingival phenotype have more pain and discomfort during oral hygiene therefore making it more difficult for plaque control.

Various techniques are used to increase the thickness of the peri-implant mucosa. These include connective tissue grafts, platelet-rich fibrin and xenogeneic collagen matrix. The volume of labial bone may be maintained by the increased thickness of soft tissue as a result of connective tissue graft . The autologous connective tissue graft has been widely recommended for mucosal tissue thickness enhancement due to its favorable thickness with minimal shrinkage in long-term follow-up when compared to other soft tissue graft approaches. Connective tissue graft (CTG) is considered the gold standard for soft-tissue correction and augmentation surgeries, but involves a secondary donor area and its associated complications. Connective tissue graft (CTG) has become a reliable treatment modality for increasing gingival thickness, width of keratinized gingiva, root coverage, treatment of furcation alveolar ridge deficiencies management of peri-implant tissue abnormalities and papillary loss. The scope of free gingival graft has been narrowed down especially in the esthetic region.

Leukocyte and Platelet rich fibrin is a second generation platelet concentrate that was introduced by choukroun et al in 2001 after platelet rich plasma. PRF is the first source of autogenous blood derived growth factors harvested without the use of anticoagulants. It is obtained by a simple and inexpensive procedure that does not require biochemical blood handling. Platelet-rich fibrin (PRF) is increasingly becoming popular in dentistry due to its growth factor-secreting properties and is also known to enhance wound healing and soft tissue thickness at the surgical site.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients between 18-60 years. 2. With thin gingival phenotype with a peri-implant mucosal thickness of less than 2mm28. With single missing tooth in the incisor, canine and premolar area. With the presence of two natural adjacent teeth and to not have a bone augmentation procedure before or during the dental implant.

  3. Patient consent approval and signing 4. Medically free patients 5. Patients with good oral hygiene 6. Patients free from untreated periodontal disease

Exclusion Criteria:

* 1. Smokers 2. Psychological problem 3. Pregnancy 4. Systemic disease 5. Poor oral hygiene 6. Patients who previously received radiation therapy of the jaws 7. Patients taking medications that affect healing.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2026-01-16 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Gingival thickness | 6 months
  Anesthetic needle with a rubber stopper36 Numerical (mm)

SECONDARY OUTCOMES:
Postoperative pain (direct) | 14 days
  Visual analogue scale.
Width of keratinized mucosa | 6 months
  Graduated periodontal probe

CONTACTS AND LOCATIONS:
Locations (1):
- The British University in Egypt, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided